CLINICAL TRIAL: NCT05932654
Title: A Phase 2a, Multicenter, Proof-of-Concept Clinical Trial to Evaluate Efficacy and Safety of BSI-045B mAb Injection in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: POC Study to Evaluate BSI-045B in Moderate-to-severe Atopic Dermatitis
Acronym: ADAMANT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSI-045B-002
Record Dates: First submitted 2023-06-05; First posted 2023-07-06 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 300 mg (Experimental): BSI-045B 300 mg SC QW × 4 weeks, then BSI-045B 300 mg SC Q2W through Week 24
  Interventions: Drug: BSI-045B

INTERVENTIONS:
Drug: BSI-045B — Patients will be treated with BSI-045B.

SUMMARY:
The study is a multicenter clinical trial and is designed as a proof-of-concept study to evaluate the efficacy, safety, tolerability, PK, immunogenicity, and PD of BSI-045B following SC injections.

The study will enroll patients with moderate to severe AD to receive the 300 mg treatment. BSI-045B wil be firstly given weekly during Week 1 to Week 4, and then every 2 weeks (Q2W) to Week 24.

DETAILED DESCRIPTION:
This study is a Phase 2a, proof-of-concept clinical study designed to evaluate the efficacy, safety, tolerability, PK, immunogenicity, and PD of BSI-045B injection in patients with moderate to severe AD. The study will be unblinded.

Following a loading dose of BSI-045B (300 mg) SC QW for 4 weeks, patients will move to maintanence 300 mg SC Q2W through Week 24. There will be a 12-week Follow-up Period after treatment.

A Safety Steering Committee (SSC) will monitor the study to identify questions concerning safety.

The primary efficacy endpoint is the proportion of patients with ≥EASI75 at Week 26 (2 weeks after last dose at Week 24), compared with baseline (Day1). Additional efficacy outcomes also include other scores on EASI, Investigator's Global Assessment (IGA), Facial IGA, and Peak Pruritus Numerical Rating Scale (PP-NRS). Efficacy assessments will be conducted at Screening, within the first hour prior to dosing on Day 1, at all subsequent visits, and at the time of early withdrawal from the study.

ELIGIBILITY:
Main inclusion Criteria:

* In the opinion of the Investigator, the patient is capable of understanding and complying with protocol requirements.
* The patient signs and dates a written ICF prior to the initiation of any study procedures.
* The patient has a diagnosis of AD (according to the criteria established by Hanifin and Rajka, 1980). The diagnosis of AD must have been present for at least 1 year, and the patient's AD must have been active for at least 3 months.
* The patient is aged 18 to 65 years, inclusive at the time of consent. Patients of any gender are eligible.
* The EASI is ≥12 at Screening and on Day 1.
* The score on the IGA is ≥3 (scale of 0 to 4) at Screening and on Day 1.
* The total body surface area (BSA) affected by AD is ≥10% as assessed by the physical examination at Screening and on Day -1.
* The patient has not received prior treatment with topical or systemic medications OR the patient has active disease despite topical or systemic treatment as per the Investigator at the time of screening.
* A male patient who is non-sterilized and sexually active with a female partner of childbearing potential, and female patient of childbearing potential who is sexually active with a non-sterilized male partner agrees to use highly effective contraception from the time of signing the ICF throughout the duration of the study and for 90 days (~5 half lives) after the last dose of study drug.

Main Exclusion Criteria:

* The patient has another dermatologic condition that might confound a diagnosis of AD or a treatment assessment.
* The patient has any clinically significant illness that may affect the safety, increase the risk for seizure or lower the seizure threshold, or potentially confound the study results.
* The patient has abnormal laboratory values during the Screening Period: ALT and/or AST > 1.5 ULN, total bilirubin ≥ 1.5 mg/dL, estimated glomerular filtration rate (GFR) < 60 mL/min (based on Cockcroft-Gault calculation), hemoglobin≤ 10 g/dL, platelet count ≤ 150 ×103/µL, creatine kinase > 2.5×ULN.
* The patient has a history of anaphylaxis following biologic therapy.
* The patient has a history of allergy to corticosteroids, diphenhydramine, hydroxyzine, cetirizine, or fexofenadine.
* The patient has a history of a clinically significant infection within 4 weeks prior to Screening.
* The patient has been diagnosed with a helminthic parasitic infection within 6 months prior to Screening.
* The patient has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to Screening or is unwilling to agree to abstain from alcohol and drugs (including cannabinoids) throughout the study.
* The patient had a major surgical or major dental procedure within 8 weeks prior to Screening.
* The patient is pregnant or lactating or intends to become pregnant or donate ova before, during, or within 90 days (~ 5 half-lives) since the last dose of study drug.
* If male, the patient intends to donate sperm during this study or within 90 days (~ 5 half-lives) since the last dose of study drug.
* The patient has a history of neurologic abnormalities including abnormal electroencephalography, brain injury including traumatic injury, perinatal cerebropathy, postnatal brain damage, blood-brain barrier abnormality, and cavernous angioma.
* The patient has a history of cerebral arteriosclerosis.
* The patient has a history of cancer. Patients with localized basal cell carcinoma, localized squamous cell carcinoma of the skin, or carcinoma in situ of the cervix may be included in the study if they have completed curative treatment at least 12 months prior to Screening. Patients with other malignant tumors may be included if they have completed curative treatment at least 5 years prior to the first dose of study drug.
* The patient has a positive test result for hepatitis B surface antigen (HbsAg), antihepatitis C virus (HCV), a history of active tuberculosis, a positive test result for human immunodeficiency virus (HIV), or a known history of HIV infection at Screening.
* The patient has poor peripheral venous access.
* The patient has donated or lost ≥ 450 mL of blood (including plasmapheresis) or had a transfusion of any blood product within 90 days prior to the first dose of study drug.
* The patient has an abnormal ECG at Screening or on Day -1. In the case of a corrected QT interval (Fridericia) (QTcF) > 450 ms or > 470 ms (patients with bundle branch block) or PR interval outside the range of 115 to 220 ms, assessment may be repeated once for eligibility determination at Screening and/or on Day -1.
* The patient has a supine systolic blood pressure < 90 or > 144 mm Hg or a supine diastolic blood pressure < 50 or > 94 mm Hg at Screening or on Day -1. If out of range, assessment may be repeated once for eligibility determination at Screening and/or on Day -1.
* The patient has a resting heart rate < 40 or > 90 bpm (not on ECGs) and considered clinically significant by the Investigator at Screening or on Day 1. If out of range, the assessment may be repeated once for eligibility determination at Screening and/or on Day -1.
* The patient plans to use any other prohibited medication or undergo any prohibited procedure during the study. Oral antibiotics are permitted. Bleach baths are not permitted.
* The patient has a risk of suicide on the Patient Health Questionnaire-2 (PH 2) or in the judgment of the Investigator, or the patient has made a suicide attempt or has a history of deliberate self-harm in the 6 months prior to Screening.
* The patient is compulsorily detained for a medical or psychiatric illness.
* The patient or their immediate family are personnel at the clinical site.
* The patient is unable to comply with restrictions and prohibited activities/treatments as listed in the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - First OC Dermatology - Fountain Valley, Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Profound Research LLC - Nashville - Corporate, Oceanside, California
  - The George Washington University School of Medicine and Health Science, Washington D.C., District of Columbia
  - Advanced Medical Research - Medical Dermatology Specialists, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - Skin Sciences/Derm Research Pllc., Louisville, Kentucky
  - Allcutis Research - Beverly, MA, Beverly, Massachusetts
  - Beacon Clinical Research, Quincy, Massachusetts
  - Sadick Research Group, New York, New York
  - Accellacare - Cary, Cary, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - Accellacare-Wilmington, Wilmington, North Carolina
  - Wright State Physicians Health Center, Fairborn, Ohio
  - Paddington Testing Company, Philadelphia, Pennsylvania
  - Center for Clinical Studies - Webster, Webster, Texas
  - Dermatology Specialists of Spokane, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
No plan.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 300 mg
Started | 22
Completed | 17
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | 300 mg
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.08 (3.536)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving at Least 75% Reduction in Eczema Area and Severity Index [EASI] at Week 26
Description: The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Time Frame: Week 26
Measure: Number (95% Confidence Interval); unit: percentage of patients achieved EASI75
Arm/Group | 300 mg
Number analyzed (Participants) | 17
percentage of patients achieved EASI75 | 94.1 [71.3 to 99.9]

2. Primary Outcome: Safety Profile of Study Treatment
Description: Number of Participants With Treatment-emergent Adverse Events
Time Frame: Day 1 to Week 36
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg
Number analyzed (Participants) | 22
Participants | 13

3. Secondary Outcome: Pharmacokinetic Parameters
Description: BSI-045B Serum Concentration
Time Frame: Weeks 4, 24, and 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 300 mg
Number analyzed (Participants) | 22
ng/mL
  serum concentration at Week 4 | 68811.694 (23168.040)
  serum concentration at Week 24 | 63876.475 (27824.166)
  serum concentration at Week 26 | 54324.171 (25546.549)

4. Secondary Outcome: Immunogenicity Following BSI-045B Treatment
Description: Number of Participants With Anti-BSI-045B Anti-drug Antibodies (ADA) Following BSI-045B Treatment
Time Frame: Day 1 to Week 36
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg
Number analyzed (Participants) | 22
Participants
  Patients with positive ADA during treatment period | 0
  Patients with positive ADA during follow-up period | 1
  Patients with positive ADA during the study | 1

5. Other Pre Specified Outcome: Exploratory Endpoint, Proportions of Patients Achieving at Least 50%, 90% Reductions in EASI
Description: as for outcome 1
Time Frame: Week 26
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Percent Change From Baseline in EASI at Each Visit
Description: as for outcome 1
Time Frame: Day 1 to Week 36
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Exploratory Endpoint, Proportion of Patients Achieving Investigator's Global Assessment (IGA) 0 or 1 at Week 26
Description: The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Day 1 to Week 36
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Exploratory Endpoint, Percentage Changes in Peak Pruritus Numerical Rating Scale (PP-NRS) at Week 26
Description: Patients will assess their worst itch severity over the past 24 hours using an 11 point NRS ('Worst Daily Pruritus NRS') with 0 indicating 'no itch' and 10 indicating 'worst itch imaginable'.
Time Frame: Day 1 to Week 36
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Proportion of Patients Achieving Facial IGA 0/1 at Week 26
Description: The facial IGA is an instrument used in clinical trials to rate the severity of the subject's facial AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Day 1 to Week 36
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory Endpoint, Conjunctivitis
Description: Occurence of conjunctivitis
Time Frame: Day 1 to Week 36
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 1 to Week 36
Arm/Group | 300 mg
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 5/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg (N=22)
headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT05932654/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT05932654/SAP_001.pdf